CLINICAL TRIAL: NCT00329940
Title: Assessment of Rheumatologic Tolerability of Letrozole in Postmenopausal Patients With Hormone Receptor Positive Breast Cancer Having Discontinued Anastrozole Adjuvant Treatment Due to Musculoskeletal Disorders
Brief Title: Safety and Rheumatologic Tolerability of Letrozole in Postmenopausal Patients With Hormone Receptor Positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345DFR04
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: Letrozole; breast cancer; critical musculoskeletal; postmenopausal; rheumatologic tolerance
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

ARMS (1):
- Letrozole (Experimental): to evaluate the rheumatological tolerability of Femara
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole
  Other Names: Femara

SUMMARY:
The purpose of this study is to assess rheumatologic tolerability of letrozole in postmenopausal patients with hormone receptor positive breast cancer having discontinued anastrozole adjuvant treatment due to musculoskeletal disorders.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women receiving anastrozole adjuvant therapy for hormone receptor positive breast cancer who want to interrupt the treatment because of severe rheumatologic adverse events
* Polymorphonuclear neutrophils (PNN) ≥ 1200/mm3, platelets ≥ 100000/mm3, hemoglobin (Hb) ≥ 10 g/dL
* Bilirubin ≤ 30 μmol, SGOT/SGPT < 3N
* Fully signed informed consent

Exclusion Criteria:

* Pain due to bone fracture
* Metastatic disease
* Hormone therapy other than anastrozole
* Incapacitating or uncontrolled concomitant disease that could hamper patient's quality of life
* Hypersensitivity to letrozole or its components

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-11; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the rheumatological tolerability of letrozole 2.5 mg/day in patients treated with anastrozole 1 mg/day | at 1, 3 and 6 months of letrozole treatment

SECONDARY OUTCOMES:
To determine the causes of discontinuation | at 1, 3 and 6 months of letrozole treatment
To determine how long letrozole treatment is maintained | at 1, 3 and 6 months of letrozole treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Saint-Cloud, France